CLINICAL TRIAL: NCT04619862
Title: Efficacy of Gabapentin in Treating Pain in Children With Severe Neurological Impairment
Brief Title: Efficacy of Gabapentin in Treating Pain in Children With SNI (Gabapentin Trial)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Child-Bright Network (Other); BC Children's Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Harold Siden, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: H20-02023
Record Dates: First submitted 2020-10-27; First posted 2020-11-06 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Pain; Neuropathic Pain; Irritability
MeSH Terms: conditions — Pain; Neuralgia | interventions — Gabapentin

STUDY DESIGN:
Intervention Model Description: This trial uses a single randomized multiple-measures cross-over design (N-of-1), with results aggregated over several subjects. In the trial, each patient will switch between gabapentin (G) and placebo (P). The sequence of whether G precedes P (GP) or P precedes G (PG) will be randomized and neither the clinician nor the subject (parent/caregiver) will know the sequence. Each subject will serve as their own control and experiment, allowing for a finer assessment of the treatment efficacy within each patient.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Both active drug and placebo will be masked in a liquid formulation, and administered via the same route (oral, direct gastric route, or direct jejunal route) depending on the subject's usual feeding approach. The label applied to the bottle will be blinded and identical flavouring will be added to the drug and placebo for additional masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Medication (Experimental): Gabapentin is clinically started at a low dose and titrated to clinical effect or maximum target dose, whichever is lower.
  The starting dose of gabapentin will be 5 mg/kg administered as oral liquid or via gastric or jejunal routes. On Day 1 of the study, the gabapentin will be administered once at bedtime and then increased according to a preset schedule. The dose will be increased every 3rd - 4th day in a step wise fashion of 13% - 50%, starting with the evening dose in order to accommodate sedation. The maximum dose for subjects will be as follows: < 15 kg to 60 mg/kg day and ≥15 kg to 45 mg/kg/day.
  Interventions: Drug: Gabapentin
- Placebo (Placebo Comparator): Participants on this arm receive placebo, masked and dispensed according to the same preset schedule as the Medication arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin — See arm descriptions
  Arms: Medication
Drug: Placebo — See arm descriptions
  Arms: Placebo

SUMMARY:
Children born with severe brain-based developmental disabilities frequently experience persistent unexplained periods of pain and irritability, often compounded by a limited capacity to communicate their distress. The investigators call this entity Pain and Irritability of Unknown Origin (PIUO). The rationale of this trial is to identify the clinical effect size of gabapentin in reducing and resolving pain in children with developmental brain disorders, specifically those with severe neurological impairment (SNI).

DETAILED DESCRIPTION:
Background

Children with SNI may experience nociceptive-inflammatory pain as a result of their specific medical condition or procedures. Often, however, it is not clear what underlies the pain behavior as there is no clear inciting noxious event. The investigators define this entity of pain without an obvious source as Pain and Irritability of Unknown Origin (PIUO).

The investigators' work to date has developed an efficient, focused clinical pathway to evaluate children with SNI for all potential sources of nociceptive-inflammatory pain. Using this approach the "unknown" element of pain in these children is reduced and a source of PIUO may be found in individual cases, increasing the potential for treatment. Nevertheless there are children, who at the end of a thorough evaluation guided by a clinical pathway, will still have PIUO. These children may benefit from adjuvant analgesics such as gabapentin.

The evidence base supporting the use of gabapentin for pain and irritability in infants and children with neurological impairment rests on case series publications describing a limited number of retrospective cases. The lack of prospective, randomized studies, even for this commonly used medication, underpins the rationale for this trial.

Objectives

The primary objective of the pilot trial is to evaluate the clinically significant difference of gabapentin to decrease pain and irritability in children with SNI, when the source of pain and irritability is attributed to neurological dysregulation (nociplastic pain), as measured by parent-reported pain scores.

The investigators will compare the gabapentin versus placebo along an escalating dose range for both individual subjects and for the group. The investigators will aggregate the results of the completed N-of-1 trials across all subjects to estimate the group level comparative effectiveness of gabapentin in reducing pain and irritability.

Outcomes from this study will help with designing larger randomized control trials, especially with sample size and power calculations. It will also provide prospective information on drug effect.

Trial Design

This trial uses a single randomized multiple-measures cross-over design (N-of-1), with results aggregated over several subjects. This design is well-suited to outcomes that are highly specific to each individual and not amenable to precise measurement across a large cohort. The heterogenous nature of pain and irritability responses in children are more likely to be personally specific and characteristic, rather than generalizable.

Subjects will switch between gabapentin (G) and placebo (P) in a randomized order. The sequence of whether G precedes P (GP) or P precedes G (PG) will be randomized by the study pharmacist, and neither the clinician nor the subject (parent/caregiver) will know the sequence. Each subject will serve as their own control and experiment, allowing for a finer assessment of the treatment efficacy within each patient.

The primary variable assessed is the child's pain score. Pain and irritability will be measured using the Non-Communicating Children's Pain Checklist - Revised (NCCPC-R) at specified intervals throughout the randomized sequence of G : P. Additional measures of parent/caregiver burden and impact on their daily function will be undertaken weekly with the PROMIS-57, a tool adapted to measure the impact of the child's pain and irritability on parental functioning. Other measures will be of usual, known side effects (e.g., sedation) and of any unexpected adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 months to 18 years with SNI (from any cause) with unexplained pain and irritability and whose cognitive or communication impairments prevent determination of pain location, cause, and type will be eligible to participate.
* Eligible children will have cognitive impairment or be non-verbal and have severe levels of disability equivalent to Gross Motor Functional Classification System (GMFCS) scores of 3, 4 or 5 as well as Communication Function Classification System (CFCS) level 4 or 5.
* Eligible children will score >3 on two scales administered via an Eligibility Screening that measures persistence and distress level the child is experiencing as well as identifies the type of pain and irritability as PIUO - with no obvious cause or explanation. The score of >3 on the scale measuring pain persistence and distress level confirms that the child is experiencing pain and irritability more than "a little" on "some days".
* The will be evidence of a comprehensive evaluation of PIUO in the child's medical history, showing no evidence for treatable sources (nociceptive-inflammatory) of pain and/or irritability symptoms.

Exclusion Criteria:

* Children not within the specified age range
* Children with communication capabilities and cognitive development to localize their pain.
* Participants whose pain and or irritability is diagnosed through completion of the PIUO Pathway during the enrollment phase of the trial.
* Patients with a known hypersensitivity/allergy to the study medication
* Patients who are actively participating in another experimental therapy study for pain and/or irritability.
* Patients who are a poor medical risk because of other systemic diseases or active uncontrolled infections.
* Patients who score A or B on the Pain Survey
* Patients who have an active source of nociceptive-inflammatory pain at the time of enrolment (e.g., post-operative pain)
* Patients with active renal disease, known renal impairment or glomerular filtration rate < 60 mL/min/1.73 m2 (if known).
* Patients with known significant hepatic impairment at the discretion of the investigator.
* Patients with clinically relevant abnormal ECG (if available) at the discretion of the investigator.
* Patients with diagnosis of sickle cell disease.
* Parents who do not speak one of Canada's two official languages (English or French)

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Mean pain and irritability score | Days 11-19
  The mean pain and irritability score on the Non-Communicating Children's Pain Checklist Revised (NCCPC-R) on active drug compared to placebo.

SECONDARY OUTCOMES:
Identification of lowest effective dose | Days 11-19 on active drug
  For patients who benefited from gabapentin, identification of the lowest dose that was effective in reducing pain scores, as shown by a lower Non-Communication Children's Pain Checklist - Revised (NCCPC-R) score compared to baseline.
Maximal effect dosage | Days 11-19 on active drug
  For patients who benefited from gabapentin, identification of the maximal effect dosage as measured by the largest improvement in the Non-Communicating Children's Pain Checklist - Revised (NCCPC-R) score compared to baseline.
Identification of latency time | Days 0-19
  Identification of the latency time in days to the onset of maximum relief of pain and irritability as measured by the Non-Communication Children's Pain Checklist - Revised (NCCPC-R) score
Adverse Events collection | Through Sequence 1 and 2, total of 55 days
  Adverse Events collection demonstrates the AEs on treatment arm do not exceed the frequency found in the Product Monograph for children receiving gabapentin

OTHER OUTCOMES:
Improvement in parent fatigue levels | Day 1 of Sequence 1 and 2 (each Sequence is 26 days with a 3 day washout period in between) and Study End, day 55
  Patient Reported Outcome Measures Information System - 57 (PROMIS-57) scores on the medication arm compared to the placebo arm

CONTACTS AND LOCATIONS:
Overall Officials: Hal Siden, MD, Principal Investigator — BC Children's Hospital Research Institute
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Optimizing the Management of Pain and Irritability in Children with Severe Neurological Impairment — http://www.paindetectives.org

DOCUMENTS (1):
  • Study Protocol (2020-10-04): https://cdn.clinicaltrials.gov/large-docs/62/NCT04619862/Prot_000.pdf